CLINICAL TRIAL: NCT00588484
Title: Determination of the Precision and Clinical Utility of Ultrasound-based Intima-Media Thickness Measurements
Brief Title: Ultrasound-based Intima-Media Thickness Measurements
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Nicholas J. Hangiandreou, Ph.D., Mayo Clinic
Other Study IDs: 2466-02
Record Dates: First submitted 2007-12-25; First posted 2008-01-08 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Carotid Artery Intima Media Thickness
Keywords: Carotid artery; Common carotid artery; Measurement; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Men, age 35 to 65, being seen at the Mayo Clinic Department of Cardiovascular Health clinic, or has an appointment for a carotid duplex ultrasound exam.
- 2: Women, age 35 to 65, being seen at the Mayo Clinic Department of Cardiovascular Health clinic, or has an appointment for a carotid duplex ultrasound exam.

SUMMARY:
Develop a standard technique and demonstrate adequate precision for measurement of intima-media thickness (IMT) for routine clinical use.

DETAILED DESCRIPTION:
IMT is measured using software to analyze ECG-gated US image sequences acquired using a standard protocol. Two sonographers acquire images and measure IMT for 100 vessels. IMT technique standard deviation (SD) is determined by assuming normally distributed measurements, and dividing the SD of the 100 (paired) IMT differences by sqrt(2). This SD will be taken as measures of precision of the IMT technique.

ELIGIBILITY:
Inclusion Criteria:

* Must have an appointment at either the Cardiovascular Health Clinic or scheduled for a carotid ultrasound.

Exclusion Criteria:

* Carotid endarterectomy,carotid stenting, carotid repair, less than 45 degree range of motion in the neck, and/or cannot lie flat on back.
* Participants Enrolled who are found after imaging not to exhibit a ~1cm long common carotid far wall region free of focal plaque in which to measure IMT will not have their data analyzed further.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 75 Men and 75 women, ages 35-65, being seen either at the Mayo Clinic Cardiovascular Clinic, or having an appointment for a carotid duplex ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2002-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary statistical endpoint for this study is to determine the standard deviation and 95% confidence interval of IMT measurements obtained using our standard method. | Four years

SECONDARY OUTCOMES:
Standard deviation and 95% confidence interval of our IMT measurement method considering data subsets with variable US image quality levels, and different levels of image plane correlation. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J. Hangiandreou, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States